CLINICAL TRIAL: NCT04828876
Title: The Effect of Yoga on Sleep and Quality of Life in Epilepsy Patients
Acronym: Yoga
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zülfünaz ÖZER (Other)
Responsible Party: Sponsor-Investigator, Zülfünaz ÖZER, PhD., Assistant Prof, Istanbul Sabahattin Zaim University
Organization: Istanbul Sabahattin Zaim University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy
Keywords: yoga; Sleep; Quality life
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups.
Who Masked: Participant
Masking Description: Yoga and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga practice (Experimental): The yoga practice will be held 2 days a week for 6 weeks, a total of 12 sessions. Each session is set as one hour
  Interventions: Behavioral: Yoga practice
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Behavioral: Yoga practice — Yoga basically consists of breathing techniques, asanas (postures) and relaxation phases.
  Practiced Yoga Stages; 10 min. standing breathing exercise, 10 min. breathing exercise with seated asana, 10 min. lying down breathing exercise with asana, 20 min. sitting breathing exercise, 10 min. The session will be completed in 60 minutes, including deep relaxation stages by lying down. At the end of each session, patients' feedback about yoga practice will be received.
  Arms: Yoga practice

SUMMARY:
Determining the sleep quality and quality of life of epilepsy patients and offering solutions can be effective in their success both in their professional and social lives.

Therefore, in this study, it was aimed to evaluate the effectiveness of yoga therapy on sleep quality and quality of life in epilepsy patients.

DETAILED DESCRIPTION:
Yoga is an ancient Hindu practice with documented therapeutic effect in western countries and means perfect control of the body, emotions and mind. It consists of breathing exercises, asanas (posture), relaxation and meditation exercises. Through breathing exercises, various postures, and meditation in yoga, the connection between mind and body is established and a balanced health is assisted.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with epilepsy for at least six months,
* Does not have any disease that causes insomnia and does not use sleeping pills
* Have not participated in a similar regular exercise program in the last 6 months,
* Seizures are under control,
* Do not have a physical illness or cognitive deficiency and a psychiatric disease that prevents understanding of the education given

Exclusion Criteria:

* Epilepsy patients who do not agree to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale in Epilepsy | 1. week
  Quality of life
Quality of Life Scale in Epilepsy | 6. week
  Quality of life

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 1. week
  Sleep
Pittsburgh Sleep Quality Index | 6. week
  Sleep

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz ÖZER, PhD, Study Chair — Istanbul Sabahattin Zaim University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozer Z, Bahcecioglu Turan G, Aksoy M. The effects of yoga on dyspnea, sleep and fatigue in chronic respiratory diseases. Complement Ther Clin Pract. 2021 May;43:101306. doi: 10.1016/j.ctcp.2021.101306. Epub 2021 Jan 19. PMID 33545575
- [Result] Amaravathi E, Ramarao NH, Raghuram N, Pradhan B. Yoga-Based Postoperative Cardiac Rehabilitation Program for Improving Quality of Life and Stress Levels: Fifth-Year Follow-up through a Randomized Controlled Trial. Int J Yoga. 2018 Jan-Apr;11(1):44-52. doi: 10.4103/ijoy.IJOY_57_16. PMID 29343930